CLINICAL TRIAL: NCT02085421
Title: Transcranial Direct Current Stimulation and Cognitive Remediation Therapy for Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSYCH-2016-23547
Record Dates: First submitted 2014-03-06; First posted 2014-03-12 (Estimated); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Psychosis
Keywords: tdcs, neuromodulation, CRT, psychosis, schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Creatine deficiency, X-linked; Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS (Active Comparator): The active tDCS will be applied at a current of 1-2mA via two saline soaked electrode sponges (3 cm x 4.5 cm) for the first 20 minutes of each CRT session in the active condition.
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): In the sham condition, tDCS will be ramped up to 1-2 mA via two saline soaked electrode sponges (3 cm x 4.5 cm) over the first 30 seconds of each CRT session and then turned off.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Transcranial direct current stimulation (tDCS) is a form of non-invasive neuromodulation that has been shown to enhance learning. tDCS is applied with current intensity of 1-2 mA of direct current and can be applied both before and during each cognitive remediation treatment session. Two saline soaked electrode sponges will be applied to the scalp.
  Other Names: transcranial direct current stimulation

SUMMARY:
The proposed pilot study is a randomized controlled study to assess effectiveness of transcranial direct current stimulation (tDCS) to enhance cognitive remediation therapy in patients with psychotic disorders. tDCS. Patients will be randomized into two arms: active tDCS vs. sham tDCS. The active tDCS will be applied at a current of 1-2 mA (milliamperes) via two saline soaked electrode sponges (3 cm x 4.5 cm) applied to the side of the head. The investigators hypothesis is that the use of tDCS will enhance the improvement seen with cognitive remediation therapy.

DETAILED DESCRIPTION:
The proposed pilot study is a randomized controlled study to assess effectiveness of tDCS to enhance cognitive remediation therapy in patients with psychotic disorders. All patients will participate in cognitive remediation therapy (CRT). After initial consent form has been signed, all participants will undergo various neurocognitive and psychological assessments including the Brief Assessment of Cognition in Schizophrenia (BACS), an EEG, and several other tasks/assessments. Participants will then complete 2-4 CRT sessions per week, each lasting approximately one hour, for a total of 10 sessions. The CRT will use a commercially available PositScience software package. Each CRT session involves an in-session assessment of skill acquisition, as collected by commercially available CRT software.

Patients will be randomized into two arms: active tDCS vs. sham tDCS. The tDCS will be applied at a current of 1-2mA via two saline soaked electrode sponges (3 cm x 4.5 cm) each CRT session. The anode will be placed over left DLPFC (dorsolateral prefrontal cortex) at F3, according to the 10-20 international system for EEG electrode placement. The cathode will be placed over the contralateral supraorbital area (Fp2). This placement is consistent with previous protocols targeting working memory. Both active and sham conditions will have identical electrode placement.

After electrodes have been placed, the participants will be instructed to log into CRT software using a unique patient identifier. Once logged in to CRT software they will be instructed to begin the session.

The tDCS will be applied at a current of 1-2mA via two saline soaked electrode sponges (3 cm x 4.5 cm) for the first 20 minutes of each CRT session in the active condition. In the sham condition, tDCS will be ramped up to 1-2 mA via two saline soaked electrode sponges (3 cm x 4.5 cm) over the first 30 seconds of each CRT session and then turned off.

Participants will complete the hour long CRT session. The software program instructs the patient when the end of the session has been reached.

At the completion of the 10 sessions of CRT, both active and sham tDCS patients will repeat the the same assessments from the beginning, including the BACS, another EEG, and several other tasks/assessments. Patients will also be asked to return for a 1-month follow-up where most of the same tasks/assessments are completed.

The consent and baseline assessments take about 8 hours in total and can be split up into 2-4 appointments. Each of the 10 training sessions lasts approximately 1 hour for a total of 10 hours of training. The post-training assessments take about 6 hours and can be split up into 2-3 appointments. The 1-month follow-up takes approxmately 3.5 hours and can be completed in 1-2 appointments. The total time commitment for this study is approximately 28-32 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Meet diagnostic criteria for schizophrenia or schizoaffective disorder
2. Are age 18-64
3. Fluent in written and spoken English
4. Have an outpatient status of at least 1 month prior to participation
5. Has been on a stable dose of psychiatric medication for at least one month prior to participation

Exclusion Criteria:

1. History of seizures or epilepsy
2. Metallic cranial plates, screws, or implanted devices
3. History of craniotomy
4. History of stroke
5. History of eczema on scalp
6. Pre-existing sores or lesions at sites of tDCS electrode placement
7. Non removable facial piercings
8. Current or possibility of current pregnancy
9. Has received a clinically meaningful dose of a targeted cognitive training intervention in the last 12 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian S Ramsay, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 18 | 15
Completed | 13 | 13
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 9 | 6 | 15
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Brief Assessment of Cognition in Schizophrenia (BACS) From Baseline to Post-Training
Description: Clinician-administered neurocognitive battery that assesses the aspects of cognition found to be most impaired and most strongly correlated with outcome in patients with schizophrenia.
  Brief Assessment of Cognition in Schizophrenia (BACS) - post training composite z-score range Arm 1 = -2.46 - 2.24 range Arm 2 = -7.67 - 0.83 Higher scores represent better cognitive performance. The BAC APP composite z-score is calculated as the sum of the subscale z-scores (i.e., verbal memory, digit sequencing, verbal fluency, symbol coding, and tower of london), adjusted by participant age and sex.
  The primary outcome measure from the BACS is a composite z score, with 0 representing the population mean, normed by age and gender.
Time Frame: Baseline, 3-5 weeks
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 13
z-score | -0.67 (1.17) | -1.68 (2.33)

2. Primary Outcome: Change in the Virtual Reality Functional Capacity Assessment Tool (VRFCAT) From Baseline to Post-Training
Description: The VRFCAT is a performance-based functional capacity measure and the 'total recipes accessed' variable represents one component of the full measure. Using a realistic virtual reality environment, the VRFCAT assesses a subject's ability to complete instrumental activities associated with a shopping trip. This provides an estimate of performance on everyday functional tasks. The summary measures include: total time (seconds), total errors, total progressions, total bus schedule checks, total recipe checks. There is no combined total score for this Tool. The minimum number of recipe checks is 0 and there is no maximum number of recipe checks for this task. A higher score on the summary measure 'total recipe checks' indicates worse performance. This means that the higher the number of times a subject consults the reference materials (i.e., recipe), the worse the performance. Based o
Time Frame: Baseline, 3-5 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 6 | 4
scores on a scale | 12.67 (1.97) | 11 (2.94)

3. Primary Outcome: Change in the D-prime Score of the N-Back Working Memory Test From Baseline to Post-Training
Description: N-back testing is a performance task used to assess working memory. In this task, pairs of numbers are presented on a computer screen, and participant are instructed to press a button whenever the pair of numbers corresponds to the pair of numbers presented two trials before (2-back). Number of hits and number of false alarms are used to calculate d-prime, the primary outcome. Depending on the number of trials completed, the range of d-prime is expected to be from -4.46 (0 hits, 80 FA) to +4.46 (20 hits, 0 FA), based on the literature. In our study, hits ranged from 3-56 and false alarms ranged from 1-146, therefore d-prime ranged from -0.42-4.02 in the full sample for the 2-back condition. A lower score on d-prime indicates worse performance.
Time Frame: Baseline, 3-5 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
units on a scale | 1.99 (1.12) | 1.42 (1.09)

4. Secondary Outcome: N-Back - Post Training 2-back Number of Hits Provided Here
Description: reflects the number of correct responses and the unit is the number of trials. Number of hits and number of false alarms are used to calculate d-prime, the primary outcome.
Time Frame: 3-5 weeks
Measure: Mean (Standard Deviation); unit: number of trials
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
number of trials | 39.88 (11.67) | 38.88 (8.41)

5. Secondary Outcome: N-Back - Post Training 2-back Number of False Alarms Provided Here
Description: reflects the number of times the participant incorrectly indicates that there is a match (when there is not) and the unit is the number of trials. Number of hits and number of false alarms are used to calculate d-prime, the primary outcome.
Time Frame: 3-5weeks
Measure: Mean (Standard Deviation); unit: number of trials
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
number of trials | 24.75 (28.05) | 49.63 (50.36)

ADVERSE EVENTS:
Time Frame: 3-5 weeks
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 11/18 | 11/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS (N=18) | Sham tDCS (N=15)
headache (General disorders) | 4 (4) | 2 (2)
neck pain (General disorders) | 0 (0) | 4 (4)
scalp pain (General disorders) | 3 (3) | 2 (2)
tingling (General disorders) | 5 (5) | 4 (4)
itching (General disorders) | 2 (2) | 3 (3)
burning sensation (General disorders) | 4 (4) | 6 (6)
skin redness (General disorders) | 0 (0) | 0 (0)
sleepiness (General disorders) | 7 (7) | 4 (4)
trouble concentration (General disorders) | 2 (2) | 3 (3)
acute mood change (General disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT02085421/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT02085421/ICF_001.pdf